CLINICAL TRIAL: NCT05092594
Title: The Prognostic Value of IgM in Covid-19 Infection
Brief Title: Prognostic Value of IgM in Covid-19 Infection
Acronym: COVID-M
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 21JGD-COVIDM
Record Dates: First submitted 2021-10-01; First posted 2021-10-25 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-03

CONDITIONS: COVID-19
Keywords: Covid-19; anti SARS-Co-V-2 IgM
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood sampling between day 1 to day 14 from first syndromes of Covid-19 infection. Serum or plasma conservations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objective of the research is to study the relation between the presence and /or the anti SARS-Co-V-2 IgM level in an early stage of COVID-19 infection, and the evolution of the illness.

DETAILED DESCRIPTION:
The secondary objective is to determinate in what manner response of IgM anti-SARS-Co-V-2 relates to patient's immunity statute, in regards to the other so-called humain "seasonal coronavirus".

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years;
* Have been diagnosed positive of SARS-CoV-2 in the Virological Laboratory of Ambroise Paré hospital;
* Have been blood sampled between 1 day and 14 days from the first clinical syndromes, and their collections of serum or plasma are conserved and accessible;
* Affiliated to the social security scheme or entitled;
* Informed and non-opposed to participating to the study.

Exclusion Criteria:

* Opposition of patient to participation to the study;
* Foreign patients under french AME scheme.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult SARS-CoV-2 positive patients who have blood sampling between 1 day and 14 days from the first clinical syndromes and their collections of serum or plasma are accessible.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-04 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Hospitalization | through study completion, an average of 1 month
  Absence of hospitalization versus hospitalization without ventilation during SARS-CoV-2 infection
Ventilation | through study completion, an average of 1 month
  Non ventilation versus ventilation during Covid-19 hospitalization

SECONDARY OUTCOMES:
Hospitalization at Ambroise Paré hospital | through study completion, an average of 1 month
  Hospitalization at Ambroise Paré hospital during SARS-CoV-2 infection
Oxygenotherapy | through study completion, an average of 1 month
  Use of high-flow oxygenotherapy
Ventilation | through study completion, an average of 1 month
  Ventilation during SARS-CoV-2 infection
Thoracic CT | through study completion, an average of 1 month
  Thoracic CT result during SARS-CoV-2 infection
Patient's vital statute | through study completion, an average of 1 month
  Death of hospitalized patients in Ambroise Paré hospital
IgM anti-SARS-Co-V-2 presence | through study completion, an average of 1 month
  IgM anti-SARS-Co-V-2 level

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Louis Gaillard, MD, PhD, Principal Investigator — Microbiological Laboratory - CHU Ambroise Paré - APHP

IPD SHARING:
Plan to Share IPD: No